CLINICAL TRIAL: NCT06276647
Title: Improving Health Outcomes and Equity by Targeting Postpartum Mothers at Highest Risk: a Pilot Randomized Control Trial
Brief Title: Improving Health Outcomes and Equity by Targeting Postpartum Mothers at Highest Risk
Acronym: HOME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Columbia University (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Elizabeth Howell, Chair, Department of Obstetrics & Gynecology, Perelman School of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 850584; R01MD016029 (NIH)
Record Dates: First submitted 2024-02-07; First posted 2024-02-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-01

CONDITIONS: Maternal Behavior; Postpartum Depression
Keywords: Postpartum
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient Education Pamphlet and Partner Sheet (Experimental): The study intervention consists of a patient education pamphlet and partner sheet (physically and virtually accessible) that will educate and prepare post-partum participants about health conditions (hypertension, diabetes, and depression), important health behaviors , physical and emotional postpartum symptoms, teach self-management skills, enhance social support, and connect post-partum participants with community resources. The education materials will provide simple actions that participants can utilize to address symptoms, realistic time frames for healing, danger signs to look out for and contact their physicians, and a list of resources for specific issues. The patient navigator will spend approximately 20 minutes with participants after enrollment, in the hospital. Following discharge, the patient navigator will contact each patient between 4 and 20 times, by phone and/or text with a research phone, to address questions and link participants to medical and community resources.
  Interventions: Behavioral: HOME
- Standard Postpartum Care (No Intervention): These patients will receive Standard postpartum care.

INTERVENTIONS:
Behavioral: HOME — The study intervention consists of a patient education pamphlet and partner sheet (physically and virtually accessible) that will educate and prepare post-partum patients. The patient navigator will explain this pamphlet at postpartum discharge, then will follow-up with the patients up to 30 days in the postpartum period.
  Arms: Patient Education Pamphlet and Partner Sheet

SUMMARY:
The goal of this educational clinical trial is to identify high-need women most at risk for poor outcomes following delivery, the problems they experience, and to create a system to improve quality of postpartum care for these high-need patients.

The main question[s] it aims to answer are:

1. How can the investigators help postpartum patients who have poor outcomes by decreasing the number of ED visits/readmissions for these patients within the first 30 days postpartum?
2. How can the investigators increase the ability of participants to "obtain needed services" and ability for patients to see their provider when they need to, in the 30-day post discharge period as one of the main pathways of unnecessary ED visits?

Participants will be put into the study group or control group. The study group will receive a pamphlet postpartum with helpful information as well as a patient navigator who the participants will be able to reach out to their first 30 days postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum patients who have delivered a baby at the Hospital of University of Pennsylvania
* Ages 18 or older
* Self-identify as Black (listed on chart)
* Speak English
* Able to read
* Other characteristics defined by our risk prediction model (algorithm)

Exclusion Criteria:

* Unable to provide informed consent
* Speaks a language other than English

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 214 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Emergency Department (ED) Visits and Readmissions | 1-30 days postpartum
  To obtain data for the primary outcome of postpartum morbidity and mortality as measured by Emergency Department (ED) visits and hospital readmissions in the 30-day post discharge period. Investigators will use chart reviews to obtain this ED/Readmission information.

SECONDARY OUTCOMES:
Ability to Obtain Needed Services | 1-30 days postpartum
  To detect the ability of participants to "obtain needed services" in the 30-day post discharge period as one of the main pathways of unnecessary ED visits. Investigators will measure this outcome by number of times patient is able to reach their doctor or healthcare provider by email, phone, or in-person.
  Investigators ask patients three weeks postpartum: "Please rate your ability to do the following on a scale of never-sometimes-often-always: Your ability to get through to the doctor's or midwife's office by phone,Your ability to speak to your provider by phone, Your ability to see your provider if you felt you needed to"
Depressive Symptoms | 1 day-6 months postpartum
  A score 11 or higher on the Edinburgh Postnatal Depression Scale (EPDS: a scale that ranges from 0-30), or suicidal ideation as indicated by the EPDS (If the answer to the question "The thought of harming myself has occurred to me" is: "Yes, quite often" or "sometimes," Higher scores indicate worse outcomes.
Depressive Symptoms | 1 day-6 months postpartum
  A score 20 or higher on the Patient Health Questionnaire (PHQ-9: scale ranges from 0-27).
  Higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States